CLINICAL TRIAL: NCT01453517
Title: Dialectical Behavior Therapy (DBT) for Post-Bariatric Patients Experiencing Weight Regain
Brief Title: A Psychological and Behavioral Intervention for Post-Bariatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karen Grothe, Principal Investigator, Assistant Professor, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10-004976
Record Dates: First submitted 2011-09-27; First posted 2011-10-18 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Obesity
Keywords: bariatric; obesity; post-surgery; intervention
MeSH Terms: conditions — Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Behavioral intervention for regain after bariatric surgery — 6 week intervention targeting dietary behavioral adherence, stress management, and distress tolerance skills to prevent weight regain
  Other Names: CBT-DBT intervention

SUMMARY:
The study is designed to test a pilot intervention for bariatric patients who are starting to regain weight after the 1st year post-surgery. Dialectical Behavior Therapy (DBT), an empirically supported therapy for Borderline Personality Disorder, has also successfully been applied to patients with substance use and binge eating problems. The purpose of this study is to develop and test a group intervention based on DBT and cognitive behavioral therapy (CBT) techniques for patients engaging in these maladaptive behaviors after surgery with co-occuring weight gain.

DETAILED DESCRIPTION:
Weight regain post bariatric surgery may be due to anatomical, physiological, or psychological and behavioral factors. One potential psychological and behavioral contributor to poor weight loss outcome following bariatric surgery may be low distress tolerance, characterized by emotional reactivity to stressors and lack of appropriate emotional regulation, and using eating, drinking, or other substances to improve mood. Recent research indicates that a subset of patients post-surgery experience challenges with subjective bulimic episodes, graze eating, and alcohol misuse; evidence for poorer excess weight loss (EWL) outcomes is associated with graze eating and uncontrolled eating behavior. This submission is for a pilot project designed to examine the impact of participation in a dialectical behavior therapy (DBT) plus cognitive behavioral therapy intervention delivered post-surgery on weight, psychological, and behavioral outcomes after Roux-en-Y gastric bypass surgery (RYGB) for patients experiencing weight regain relapse with co-occuring disordered eating or substance misuse behaviors.

ELIGIBILITY:
Inclusion criteria

* regained ≥ 15% of total post-surgical weight lost
* has either disregulated eating, drinking, or misuse of chemical substance
* age 18-75
* ability to participate in group
* completed first Roux-en-Y gastric bypass procedure at Mayo Clinic

Exclusion criteria

* patients with an uncontrolled psychiatric diagnosis
* patients severely impaired by drug or alcohol use
* completed surgical intervention at location other than Mayo Clinic
* more than one bariatric procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
change in weight and BMI | weighed at baseline and six weeks [weighed weekly during 6 week intervention]

SECONDARY OUTCOMES:
distress tolerance | baseline, posttreatment (within 2 weeks of intervention completion) [measured over an average of 10-12 weeks]
  emotion regulation and distress tolerance(Distress Tolerance Scale)
Mood | baseline, weekly during 6-week intervention, posttreatment (within 2 weeks of intervention completion)[measured over an average of 10-12 weeks]
  Baseline and posttreatment measure: Structured Clinical Interview for DSM Disorders (SCID)-I Mood Module) Weekly during 6-week intervention: Beck Depression Inventory II
Maladaptive eating and purging | baseline, weekly during 6-week intervention, posttreatment (within 2 weeks of intervention completion)[measured over an average of 10-12 weeks]
  Baseline and posttreatment measures: Eating Disorder Diagnostic Scale, modified Eating Disorder Examination-Q Weekly during 6-week intervention: modified Eating Disorder Examination-Q, food diary, number of eating episodes and number of snacks to quantify graze eating
Alcohol consumption | Baseline, weekly during 6-week intervention,posttreatment (within 2 weeks of intervention completion) [measured over an average of 10-12 weeks]
  Baseline: SCID-I Substance Module Weekly during 6-week intervention: quantity, frequency, type of substance use

CONTACTS AND LOCATIONS:
Overall Officials: Karen Grothe, PhD, LP, Principal Investigator — Mayo Clinic; Susan Himes, PhD, Principal Investigator — Lifespan/Brown Medical School
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States